CLINICAL TRIAL: NCT04217837
Title: Neurostar Transcranial Magnetic Stimulation (TMS) Advanced Therapy System: Data Management, Analysis, and Reporting Format for Clinical Treatment Utilization and Outcomes in the UK
Brief Title: Treatment of Major Depressive Disorder in the UK Using TMS Therapy
Status: Withdrawn | Type: Observational
Why Stopped: COVID
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Other Study IDs: 44-50011-000
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation; Major Depressive Disorder; MDD; TMS; NeuroStar Advanced Therapy System; Repetitive Transcranial Magnetic Stimulation; rTMS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Major Depressive Disorder: Participants who meet the DSM-5 clinical diagnostic criteria, in the opinion of the treating clinician, for primary diagnosis of unipolar, non-psychotic MDD.
  Interventions: Device: Transcranial Magnetic Stimulator

INTERVENTIONS:
Device: Transcranial Magnetic Stimulator — Transcranial magnetic stimulation (TMS) uses a targeted pulsed magnetic field, similar to what is used in an MRI (magnetic resonance imaging) machine. While the patient is awake and alert, NeuroStar TMS Therapy stimulates areas of the brain that are underactive in depression.
  Other Names: TMS Therapy; Neurostar

SUMMARY:
The major objective of this observational study is to describe clinical outcomes of patients in the UK receiving treatment with the NeuroStar TMS Therapy system in routine clinical practice.

DETAILED DESCRIPTION:
This is a single-center, naturalistic, observational study following the use of the NeuroStar® Advanced Therapy System and assessment of clinical outcome. The goal is to collect, analyze and report information as aggregated summaries on participants receiving treatment with the NeuroStar® Advanced Therapy System.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, age 22 - 70, out-patient
2. Participants who meet the DSM-5 clinical diagnostic criteria, in the opinion of the treating clinician, for primary diagnosis of unipolar, non-psychotic MDD. The intended treatment plan uses the labeled treatment parameters for TMS as described in the NeuroStar® System
3. Women of child bearing potential must be using a medically accepted reliable means of contraception (for oral contraceptive medication: must be in use for at least 3 months)
4. Women of childbearing potential must have a negative pregnancy test at screening using urine dipstick
5. Participants must have the capacity to consent to all tests and examinations required by the protocol and must sign a written informed consent document to participate in the study.

Exclusion Criteria:

1. History of seizures or increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure or history of significant head trauma with loss of consciousness for ≥ 5 minutes
2. Inability to locate and quantify a motor threshold as defined in the protocol
3. Conductive, ferromagnetic, or other magnetic-sensitive metals implanted in the participant's head within 30 cm of the treatment coil excluding the mouth that cannot safely be removed. Examples include: cochlear implants; implanted electrodes/stimulators; aneurysm clips or coils; stents; bullet fragments; jewelry; and hair barrettes
4. Any psychiatric disorder which, in the judgement of the Investigator, may hinder the participant from completing the procedures required by the study protocol
5. Active or inactive implants (including device leads), including deep brain stimulators, and vagus nerve stimulators
6. Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease
7. Known or suspected pregnancy

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical Practice
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression - Severity Scale | Baseline, 6 weeks, 3, 6, 9, and 12 months
  The change from baseline to endpoint on the total score for the Clinical Global Impression - Severity scale will be reported for the 6 week 3, 6, 9, and 12 month time points. The 7-point scale requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The scale ranges from 1-7, where a higher score means a worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9-item Self Report | Baseline, 6 weeks, 3, 6, 9, and 12 months
  The change from baseline to endpoint on the total score for the PHQ-9 will be reported for the 6 week, 3, 6, 9, and 12 month time points. The questionnaire assesses degree of depression severity. The scale ranges from total scores of 1-27, where a higher score means a worse outcome.
Inventory of Depressive Symptomatology - Self Report (IDS-SR) | Baseline, 6 weeks, 3, 6, 9, and 12 months
  The change from baseline to endpoint on the total score for the Inventory of Depressive Symptomatology - Self Report will be reported for the 6 week, 3, 6, 9, and 12 month time points. It is a tool designed to screen for depression and measure changes in severity of symptoms. The scale ranges from total score ranges of 0-84, where a higher score means a worse outcome.
EuroQol 5 Dimensions | Baseline, 6 weeks, 3, 6, 9, and 12 months
  The change from baseline to endpoint on the total score for the EuroQol 5 Dimensions will be reported for the 6 week, 3, 6, 9, and 12 month time points. The EuroQol 5 Dimensions questionnaire assesses quality of life and is presented as a health profile.
Health Resource Utilization Questionnaire (HRU) | Baseline, 6 weeks, 3, 6, 9, and 12 months
  The change from baseline in health care service utilization reported on the individual questions contained in the HRU will be reported for the 6 week, 3, 6, 9, and 12 month time points. It is a socioeconomic and quality of life questionnaire. Because changes in individual questions are reported, there is no range of scores. The score ranges from 0-100, where a higher score means a better outcome.
Short Form 36-item Questionnaire | Baseline, 6 weeks, 3, 6, 9, and 12 months
  The change from baseline to endpoint on the Individual Factor Scores and General Medical and Mental Health Composite Scores for the SF-36 will be reported for the 6 week, 3, 6, 9, and 12 month time points. The Short Form 36-item Questionnaire evaluates quality of life outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelghani, MBBCh, MSc, MRCPsych, Principal Investigator — St. Pancras Hospital
Locations (1):
- St Pancras Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No